CLINICAL TRIAL: NCT04585334
Title: A Double Blind, Double Dummy, Multicenter, Randomized, Placebo- and Active-controlled Clinical Trial to Evaluate Effectiveness of Tricortin 1000 in Patients Affected by Chronic Low Back Pain
Brief Title: Effectiveness of Tricortin 1000 in Patients Affected by Chronic Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQ06.17.01
Record Dates: First submitted 2020-03-02; First posted 2020-10-14 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain, Mechanical
Keywords: Chronic; Degenerative process of disc and facet
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: PAES, double blind, double dummy, multicenter, randomized, controlled clinical study
Who Masked: Participant, Investigator
Masking Description: Double blind, double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A Tricortin (Experimental): Tricortin 1000 by intramuscular route
  Interventions: Drug: Tricortin 1000
- Arm B Itami (Active Comparator): Itami Diclofenac sodium medicated plaster by topical application
  Interventions: Drug: Itami
- Arm C Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tricortin 1000 — Tricortin 1000 [2 mL ampoules containing 12 mg of phospholipids and 1 mg of Vitamin B12 (Cyanocobalamin)] will be administered intramuscular on the gluteus, once daily (24 hours apart), for 15 days starting from the evening of Day 0 (visit 2) plus Diclofenac sodium medicated plaster placebo will be applied twice daily (12 hours apart) for 15 days starting from the evening of Day 0 (visit 2), i.e. 30 applications.
  Other Names: Tricortin
  Arms: Arm A Tricortin
Drug: Itami — Diclofenac sodium 140 mg medicated plaster (Itami®) will be applied twice daily (12 hours apart) for 15 days starting from the evening of Day 0 (visit 2), i.e. 30 applications plus Tricortin 1000 placebo (2 mL ampoules) will be administered intramuscular on the gluteus, once daily (24 hours apart), for 15 days starting from the evening of Day 0 (visit 2).
  Other Names: Diclofenac sodium 140 mg medicated plaster
  Arms: Arm B Itami
Drug: Placebo — Tricortin 1000 placebo (2 mL ampoules) will be administered intramuscular on the gluteus, once daily (24 hours apart), for 15 days starting from the evening of Day 0 (visit 2) plus Diclofenac sodium medicated plaster placebo will be applied twice daily (12 hours apart) for 15 days starting from the evening of Day 0 (visit 2), i.e. 30 applications.
  Other Names: Placebo plaster and Tricortin placebo
  Arms: Arm C Placebo

SUMMARY:
PAES, double blind, double dummy, multicenter, randomized, controlled clinical study to demonstrate superiority of Tricortin 1000 over placebo in improvement in pain relief as change from baseline to 15 days in patients with chronic low back pain (LBP).

DETAILED DESCRIPTION:
This is a PAES, double blind, double dummy, multicenter, randomized, controlled clinical study, which will consist of a Screening phase (Visit 1) of up to 14 days and a Follow-up phase of up to 15 days.

A total of 300 patients of either sex, aged between 40 and 70 years with diagnosis of chronic mechanical (mild, moderate degenerative process of disc and facet) LBP for at least 3 months but no more than 6 months will be randomized.

Two stratification groups will be distinguished: the first group will be comprised of patients with chronic mechanical LBP due to mild, moderate degenerative process of disc and facet from 40 to <55 years, the second group will be comprised of patients with chronic mechanical LBP due to mild-moderate degenerative process of disc and facet ≥55 to 70 years.

All patients will be required to have diagnosis of chronic LBP with clinically and imaging confirmation of mechanical (mild, moderate degenerative process of disc and facet).

Baseline assessments include: pain assessment and functional disability, clinical parameters, patient global assessment (PGA), clinical global impression (CGI) and consumption of rescue medication.

Eligible patients will then be randomly assigned to one of the following three treatment arms:

1. Tricortin 1000 by intramuscular route (Arm A)
2. Diclofenac sodium medicated plaster by topical application (Arm B)
3. Placebo (Arm C) In arm A and B, Tricortin 1000 and Diclofenac sodium medicated plaster will be administered together with the alternate placebo, while patients in the placebo arm (Arm C) will be treated with both intramuscular and locally applied placebo.

Patients will be in the study for approximately 30 days of trial duration with a treatment period of 15 days.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of mechanical (mild, moderate degenerative process of disc and facet) chronic LBP, for at least 3 months but no more than 6 months, confirmed (thanks to instrumental analysis obtained within 9 months before the Screening visit) by CT or MRI. In case a MRI/CT performed in the previous 9 months is not available, the diagnosis should be confirmed by means of a MRI performed between Screening visit (Visit 1) and Baseline visit (Visit 2)
2. A moderate to severe acute exacerbation of Chronic LBP at study entry, defined as a score ≥4 and ≤8 rated on the NRS-11
3. Age greater than or equal to 40 and less than or equal to 70 years
4. Patient able to maintain a Diary during the study
5. Patient with a Body Mass Index (BMI) < 30 kg/m2
6. Discontinuation of any analgesic/NSAID therapy, opioids, corticosteroids, skeletal muscle relaxants and any other medication or non-pharmacological therapy (if it would interfere with the study assessments), with no intent to resume during study
7. Patients who did not receive antidepressant medications and/or benzodiazepines for at least 60 days
8. Patient able to read and understand the language and content of the study material, understand the requirements for follow-up visits, is willing to provide information at the scheduled evaluations and is willing and able to comply with the study requirements
9. Patient has undergone the informed consent process and has signed an approved consent form
10. If female, patient must have a negative urine pregnancy test and use a highly effective form of contraception for at least one month prior to screening and throughout the study; or females must be surgically sterile, or postmenopausal as documented in medical history for at least one year. Highly effective birth control methods include: combined hormonal contraception (containing estrogen and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence*
11. Patients who did not use Tricortin 1000 in the past to treat LBP or other pathological conditions.

    * Note: According to 4.1 paragraph "Birth control methods which may be considered as highly effective" of the CTFG/Recommendations related to contraception and pregnancy testing in clinical trials

Baseline Inclusion Criteria:

1. In aptients for which a MRI/CT performed in the previous 9 months is not available, the diagnosis of chronic LBP should be confirmed by means of a MRI performed between screening visit (Visit 1) and baseline (Visit 2)
2. LBP with score ≥ 5 and ≤ 8 in the NRS-11 (off medication except for paracetamol, study rescue medication)
3. Patient has discontinued use of all analgesic/NSAIDs, opioids, corticosteroids, skeletal muscle relaxants, and any other medication or non-pharmacological therapy (if it would interfere with the study assessments) at V1 (except for patients that will perform the MRI between Screening and Baseline visit) and agree not to resume them during study (except for paracetamol, study rescue medication). These medication must be discontinued for at least 14 days before the Baseline visit (Visit 2/ Day 0), i.e. can be taken for maximum 7 days during the 14-21 days of Screening phase, in case that the screening phase is prolonged up to 21 days in patients that will perform the MRI between screening and baseline visit.
4. Patient has complied with the requirements for rescue medication (no more than 4 tablets - 2 grams - of paracetamol per day up to 4 days per week) and no paracetamol intake in the 24 hours before baseline visit
5. Patient continues to meet all Screening inclusion/exclusion criteria at the Baseline visit, with the exception of screening inclusion criterion 2 which is replaced by baseline inclusion criterion 2

Exclusion Criteria:

Related to patients

1. Patients suffering of chronic non-specific LBP
2. Females who are pregnant or breast-feeding
3. Patients who are not able to give informed consent
4. Patients who cannot commit to the entire duration of the study
5. Patients with back pain referred from a mechanical cause (except for mild, moderate degenerative process of disc and facet) non spinal source or back pain associated with another specific spinal cause
6. Patients who have a primary bone disease, cancer, infection (except for osteoporosis patients without fracture history)
7. Other conditions which may confound the interpretation of the study, such as carpal, rheumatoid arthritis, severe venous diseases, peripheral arterial diseases, transient ischemic attack, stroke, current symptoms of coronary artery disease
8. History of narcotic abuse at any time in the past and/or drug or alcohol abuse in the past year
9. Patients who have had a previous treatment with physical therapy for LBP in the last 4 weeks before the screening visit or are going through a course of physical therapy or chiropractic treatment at the time of planned enrolment
10. Participation in another research study
11. History of epilepsy
12. Patients who have an unstable psychiatric condition

    Red flags as possible indicators of serious spinal pathology:
13. Unexplained serious thoracic pain
14. Any recent trauma, which may raise the possibility of a fracture
15. Fever and unexplained weight loss
16. Bladder or bowel dysfunction
17. History of carcinoma
18. Progressive neurological deficit
19. Disturbed gait, saddle anaesthesia Musculoskeletal related
20. Radicular syndromes of idiopathic,metabolic, toxic, infective, demyelinating or neoplastic aetiology
21. Patients with spondylolisthesis, spondylolysis or ankylosing spondylitis.
22. Patients with scoliosis of 15° or more
23. Patients with inflammatory arthritis or severe degenerative process of disc and facet
24. Patients who have had prior spine surgery, including rhizotomy as like as, patients who are planning or have been advised to have spine surgery.

    Concomitant conditions, diseases, medications and/or clinical history
25. Patients with any concomitant chronic disease(s) or condition(s) that may predispose them to a high probability of interfering with the completion of the follow-up of the study such as peptic ulcer, liver disease, severe coronary disease, renal disease, cancer, pregnancy, alcoholism, mental state, or other clinically significant condition
26. Patients with history of active or suspected oesophageal, gastric, pyloric channel, or duodenal ulceration or bleeding in the last 12 weeks before the screening visit
27. Patients requiring chronic use of analgesia for pain
28. Patients with known allergies or hypersensitivity or intolerance to Tricortin 1000, NSAIDs and/or paracetamol, and/or to active or inactive excipients of formulation
29. Patients in treatment with neuroleptics (antipsychotics)
30. Patients affected by diabetic neuropathy, multiple sclerosis or Amyotrophic Lateral Sclerosis
31. Any contraindications to either prone distraction or side posture manipulation
32. Any contraindications as reported in the Patient Information Leaflet of Tricortin 1000 or Diclofenac sodium medicated plaster.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 15 days in patients with chronic low back pain (LBP) and acute exacerbation at study entry using Numerical Rating Scale for pain | Day 15
  The primary efficacy endpoint will be the change from baseline to Day 15 in NRS-11 score.(0-10 points Numerical Rating Scale for pain, where score 0 corresponds to no pain and score 10 corresponds to unimaginable pain)

SECONDARY OUTCOMES:
Improvement in pain relief as change from baseline to 15 days in patients with chronic LBP and acute exacerbation at study entry, using Numerical Rating Scale for pain | Day 15
  To compare Tricortin 1000 and diclofenac sodium medicated plaster (Itami®) in improvement in pain relief as change from baseline to 15 days in patients with LBP. (0-10 points Numerical Rating Scale for pain, where score 0 corresponds to no pain and score 10 corresponds to unimaginable pain)
Functional disability improvement as change from baseline to 15 days through the Oswestry Low Back Pain Disability Index (ODI), version 2.1a | Day 0, Day 7 and Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster (Itami®) in functional disability improvement. LBP related disability improvement will be measured through the Oswestry Low Back Pain Disability Index (ODI), version 2.1a, at baseline visit and then in the following visits: V3-Day 7 and V4-Day 15.
Clinical improvement as change from baseline to 15 days | Day 0, Day7 and Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster (Itami®) in clinical improvement as change from baseline to 15 days. Clinical improvement will be evaluated at baseline visit and then at V3-Day 7 and V4-Day 15 through the following parameters: Range of Motion testing, Joint reflex changes (ROT), Lasegue's test (passive straight leg raise), Femoral stretch test (Wasserman test), Dandy's sign, Valleix's points pressure.
Patient global assessment PGA as change from baseline to 15 days. PGA:single-item measure:Considering all the ways that your LBP affect you,select one response for how you are doing at the moment:0=very well;1=well;2=fair;3=poor;4=very poor | Day 0, Day7 and Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster (Itami®) in patient global assessment (PGA) as change from baseline to 15 days. PGA will be evaluated at baseline visit and then in the following visits: V3-Day 7 and V4-Day 15
ClinicalGlobalImpression as change from baseline to15days.CGI:7point scale clinician-rated(severity of illness)from1(normal)to7(severely ill).CGI score from1(very much improved)to7(very much worse).Treatment response consider efficacy and AEs | Day 0, Day7 and Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster (Itami®) in clinical global impression CGI as change from baseline to 15 days. CGI will be evaluated at baseline visit and then in the following visits: V3-Day 7 and V4-Day 15
Consumption of rescue medication as change from baseline to 15 days using a patient diary (maximum 4 tablets for 4 days/week) | From Day -14 to Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster (Itami®) in consumption of rescue medication as change from baseline to 15 days. Daily rescue medication required for pain relief up to V4-Day 15 using a patient diary
Safety as change from baseline to 15 days evaluated by physical examination (body areas:Head;Ears;Eyes;Nose;Mouth;Skin;Heart;Lung;Lymph nodes;Genitourinary;Gastrointestinal;Skeletal;Neurological systems;Other, specify) | From Day -14 to Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster in patient safety as change from baseline to 15 days.
Safety as change from baseline to 15 days evaluated by vital signs (systolic blood pressure, diastolic blood pressure, heart rate) | From Day -14 to Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster in patient safety as change from baseline to 15 days.
Safety as change from baseline to 15 days evaluated by tracking the number of patient withdrawals and their adverse events | From Day -14 to Day 15
  To compare Tricortin 1000 with placebo and diclofenac sodium medicated plaster in patient safety as change from baseline to 15 days.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (13):
- Italy (13):
  - ATS Insubria, Porlezza, Como
  - ATS Insubria, Alzate Brianza
  - UOC Medicina Fisica e Riabilitazione - Unità Spinale Unipolare, Azienda OU "Consorziale Policlinico" Bari, Bari
  - Servizio di Medicina Fisica e Riabilitativa, AOU Policlinico-P.O.G. Rodolico, Catania
  - U.O. Medicina Fisica e Riabilitativa Azienda ospedaliera Mater Domini, Catanzaro
  - ATS Insubria, Como
  - ATS Insubria, Erba
  - SODC-Riabilitazione Azienda ospedaliero-Universitaria Careggi- Ospedale Careggi, Florence
  - U.O.C. di Riabilitazione Ortopedica, Azienda Ospedaliera Universitaria di Padova, Padua
  - U.O.C. di Riabilitazione AOU Policlinico P. Giaccone, Palermo
  - U.O.C. Medicina Fisica Riabilitativa Azienda Policlinoc Umberto I, Università di Roma La Sapienza, Roma
  - UOS Medicina Fisica e Riabilitativa Azienda Ospedaliero Universitaria Sant'Andrea-Roma, Roma
  - U.O.C. Neuroriabilitazione, Dipartimento di Neuroscienze, Azienda Ospedaliera Universitaria Integrata di Verona, Policlinico Borgo Roma, Verona

IPD SHARING:
Plan to Share IPD: No